CLINICAL TRIAL: NCT02173262
Title: Feasibility of Using an Integrated Consent Model to Compare Two Standard of Care Regimens for Primary Prophylaxis of Taxotere/Cyclophosphamide-Induces Febrile Neutropenia
Brief Title: REaCT Integrated Consent Model to Compare Two Standard of Care Regimens
Acronym: OTT14-03
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20140380-01H
Record Dates: First submitted 2014-06-16; First posted 2014-06-24 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — Granulocyte Colony-Stimulating Factor; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- G-CSF (Other): Participants will receive a daily injection of G-CSF while on chemotherapy for prevention of febrile neutropenia.
  Interventions: Drug: G-CSF
- Ciprofloxacin (Other): Participants will receive Ciprofloxacin 500 mg twice a day by mouth for 10 days of each cycle during chemotherapy for prevention of febrile neutropenia.
  Interventions: Drug: Ciprofloxacin

INTERVENTIONS:
Drug: G-CSF
  Other Names: granulocyte-colony stimulating factor
  Arms: G-CSF
Drug: Ciprofloxacin
  Other Names: Cipro; Cipro XR; Proquin XR
  Arms: Ciprofloxacin

SUMMARY:
The Integrated Consent Model is being increasingly used internationally to improve patient care. In this feasibility study we will explore whether the model is feasible in practice; and whether it can be used to increase the number of physicians and patients who take part in clinical trials, and address the critical issue around the optimal febrile neutropenia prevention by randomizing eligible patients to either G-CSF or ciprofloxacin.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed primary breast cancer
* Planned TC chemotherapy
* ≥19 years of age
* Able to provide verbal consent
* Willing to complete a survey

Exclusion Criteria:

• Contraindication to either Ciprofloxacin or G-CSF

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Actual)
Dates: Start 2014-08; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The percentage of randomized patients in each physician's practice | every 4 weeks up to 2 years
  The percentage of randomized patients will be measured by collecting reasons for NOT complying with, or "opting-out" of the randomized selection compared to the overall accrual.

SECONDARY OUTCOMES:
rates of febrile neutropenia | Once when the last participant completes chemotherapy up to year 2
  Rates of febrile neutropenia will be compared between Ciprofloxacin and G-CSF

CONTACTS AND LOCATIONS:
Overall Officials: Mark Clemons, Doctor, Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Clemons M, Mazzarello S, Hilton J, Joy A, Price-Hiller J, Zhu X, Verma S, Kehoe A, Ibrahim MF, Sienkiewicz M, Stober C, Vandermeer L, Hutton B, Mallick R, Fergusson D. Feasibility of using a pragmatic trials model to compare two primary febrile neutropenia prophylaxis regimens (ciprofloxacin versus G-CSF) in patients receiving docetaxel-cyclophosphamide chemotherapy for breast cancer (REaCT-TC). Support Care Cancer. 2019 Apr;27(4):1345-1354. doi: 10.1007/s00520-018-4408-6. Epub 2018 Aug 11. PMID 30099602